CLINICAL TRIAL: NCT03676790
Title: Effect of Ultrasound Associated to Exercises in Patients With Knee Osteoarthritis
Brief Title: Ultrasound and Exercises in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Raquel A. Casarotto, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAAE: 47955315.7.0000.0065
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, Knee; Ultrasonic Therapy; Exercise Therapy; Randomized controlled trial.
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group I (Experimental): (in the first month, continuous ultrasound was applied three times a week and in the second month patients performed only exercise sessions three times a week)
  Interventions: Other: Group I
- Group II (Experimental): (in the first month, pulsed ultrasound was applied three times a week and in the second month patients performed only exercise sessions three times a week)
  Interventions: Other: Group II
- Group III (Experimental): (in the first month, the continuous ultrasound was applied three times a week and in the second month, three times a week, the continuous ultrasound associated with exercises was applied)
  Interventions: Other: Group III
- Group IV (Experimental): (in the first month, the pulsed ultrasound was applied three times a week and in the second month, three times a week, the pulsed ultrasound associated with exercises was applied)
  Interventions: Other: Group IV
- Group V (Experimental): (patients received only exercise sessions three times a week for eight weeks)
  Interventions: Other: Group V

INTERVENTIONS:
Other: Group I — Group I In the first month, continuous ultrasound was applied three times a week. In the second month, patients performed only exercise sessions three times a week. In the ultrasound treatment, the following parameters were used: frequency of 1 MHz, intensity of 1.5 W/cm2 (temporal and spatial mean SATA), duty cycle of 100%, with application time of 5 minutes on the medial side and 5 minutes on lateral side of knee.
  Exercises
  The intervention was divided into three phases: P-1, P-2 and P-3 during eight weeks with three sessions a week. Each session lasted 45 minutes:
  * 10 minutes warming-up (treadmill, ergometer bike or rowing machine);
  * 30 minutes 2-3 sets with P-1, P-2 or P-3;
  * 5 minutes stretching (hamstrings, quadriceps, adductors, and gastrocmenius).
  Arms: Group I
Other: Group II — Group II In the first month, pulsed ultrasound was applied three times a week. In the second month, patients performed only exercise sessions three times a week. In the treatment with the US, the following parameters were used: 1 MHz frequency, 2.5 w / cm2 intensity (temporal and spatial mean SATA), pulsed mode (25%), 5 minutes on the medial side and 5 minutes on the lateral side of the knee.
  Exercises
  The intervention was divided into three phases: P-1, P-2 and P-3 during eight weeks with three sessions a week. Each session lasted 45 minutes:
  * 10 minutes warming-up (treadmill, ergometer bike or rowing machine);
  * 30 minutes 2-3 sets with P-1, P-2 or P-3;
  * 5 minutes stretching (hamstrings, quadriceps, adductors, and gastrocmenius).
  Arms: Group II
Other: Group III — Group III In the first month, the continuous ultrasound was applied 3 times a week. In the second month, 3 times a week, the continuous ultrasound was applied associated with exercises. The parameters were used: frequency of 1 MHz, intensity of 1.5 w / cm2 (temporal and spatial mean SATA), continuous mode (100%), with application time of 5 minutes on the medial side and 5 minutes on lateral side of knee.
  Exercises
  The intervention was divided into three phases: P-1, P-2 and P-3 during eight weeks with three sessions a week. Each session lasted 45 minutes:
  * 10 minutes warming-up (treadmill, ergometer bike or rowing machine);
  * 30 minutes 2-3 sets with P-1, P-2 or P-3;
  * 5 minutes stretching (hamstrings, quadriceps, adductors, and gastrocmenius).
  Arms: Group III
Other: Group IV — Group IV In the first month, the pulsed ultrasound was applied three times a week. In the second month, three times a week, the pulsed ultrasound associated with exercises was applied. In the treatment with the US, the following parameters were used: 1 MHz frequency, 2.5 w / cm2 intensity (temporal and spatial mean SATA), pulsed mode (25%), 5 minutes on the medial side and 5 Minutes on the lateral side of the knee.
  Exercises
  The intervention was divided into three phases: P-1, P-2 and P-3 during eight weeks with three sessions a week. Each session lasted 45 minutes:
  * 10 minutes warming-up (treadmill, ergometer bike or rowing machine);
  * 30 minutes 2-3 sets with P-1, P-2 or P-3;
  * 5 minutes stretching (hamstrings, quadriceps, adductors, and gastrocmenius).
  Arms: Group IV
Other: Group V — Group V Patients received only exercise sessions three times a week for two months.
  Exercises
  The intervention was divided into three phases: P-1, P-2 and P-3 during eight weeks with three sessions a week. Each session lasted 45 minutes:
  * 10 minutes warming-up (treadmill, ergometer bike or rowing machine);
  * 30 minutes 2-3 sets with P-1, P-2 or P-3;
  * 5 minutes stretching (hamstrings, quadriceps, adductors, and gastrocmenius).
  Arms: Group V

SUMMARY:
The aim of this investigation is to compare the effects of continuous (CUS) and pulsed (PUS) ultrasound associated with a program of exercises on pain, range of motion, muscle strength, functionality, mobility and activity in patients with knee osteoarthritis. Participants were randomized into five groups: Group I (in the first month, continuous ultrasound was applied), Group II (in the first month, pulsed ultrasound was applied), Group III (in the first and second month, the continuous ultrasound was applied), Group IV (in the first and second month, the pulsed ultrasound was applied) and Group V (patients received only exercise sessions for eight weeks).

DETAILED DESCRIPTION:
Strong evidence suggests that joint exercises reduce pain and disability in patients with osteoarthritis. There is evidence that exercise is responsible for muscular strengthening and better flexibility, improved global function as well as better performance in activities of daily living (ADL).

There are two modes of US, continuous and pulsed. Continuous US (CUS) generates thermal effects by stimulating the process of tissue regeneration, changing cell membrane permeability and increasing intracellular calcium, while pulsed US (PUS) mainly produces non-thermal effects to increase tissue metabolism, enhance fibrous tissue extensibility and elevate pain threshold

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, participants needed to suffer knee osteoarthritis with osteoarthritis levels 2 - 4 according to Kellgren-Lawrence grade12, be aged between 50 and 75 years and suffer knee pain and functional disability for at least three months, according to the criteria of the American College for Rheumatology (ACR)13. Participants from both genders were included. The Kellgren and Lawrence grading of knee osteoarthritis is as follows: none (0), doubtful (1), minimal (2), moderate (3) and severe (4).

The ACR criteria of knee osteoarthritis are as follows:

* Using history and physical examination: knee pain and three of the following - over 50 years old; less than 30 minutes of morning stiffness; bone tenderness; bone enlargement; no palpable warmth of synovial.
* Using history, physical examination and radiographic findings: knee pain and one of the following - over 50 years old; less than 30 minutes of morning stiffness; crepitus on active motion; and osteophytes.
* Using history, physical examination and laboratory findings: knee pain and five of the following - over 50 years old; less than 30 minutes of morning stiffness; bone tenderness; bone enlargement; no palpable warmth of synovial; crepitus on active motion; ESR <40 mm/h; rheumatoid factor <1: 40; synovial fluid sign of osteoarthritis.

Exclusion Criteria:

* Participants were excluded if they had cancer, diabetes, symptomatic hip osteoarthritis, or used antidepressants, anti-inflammatory medications or anxiolytics during six months prior to enrollment.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Measure | eight weeks
  Pain was assessed using a visual analogue scale (VAS)14 consisting of a 10 cm rule (without numbers). At the left side, 'no pain' is written, while on the right side, 'unbearable pain'. Patients were instructed to mark on the rule what their level of pain was.

SECONDARY OUTCOMES:
Functionality Measure | eight weeks
  Functionality was measured using the Lequesne questionnaire,14 which consists of 11 questions about pain, discomfort and function. Scores range from 0 to 24 (from 'no' to 'extremely severe' dysfunction).
Range of motion | eight weeks
  Range of motion for flexion of the knees was measured with the universal goniometer (AESCULAP), according to the methods described by Marques.
Muscular strength | eight weeks
  Muscular strength was estimated at maximal isometric force for the quadriceps, using a portable dynamometer (Lafayette, USA). Under stabilized conditions, patients, sitting with knees flexed at 10o, 60o and 90o (measured by a goniometer),16 were asked to extend the legs as far as they could. Three trials were conducted and the mean value was obtained.
Activity | eight weeks
  Activity was measured using the Western Ontario and McMaster Universities Osteoarthritis (WOMAC) questionnaire,17 which is self-administered and measures pain, frozen joints and physical activity. Increased scores indicate decreased activity.
Mobility and balance | eight weeks
  Mobility and balance are evaluated by Timed Get Up and Go (TGUG)18 and 8 meters Test19. The TGUG quantifies in seconds the functional mobility through the time that the individual needs to perform the task of getting up from a chair, walking three meters, turning back towards the chair and sitting again. The 8-meter test measures the time and number of steps required for a person to walk for 8 meters.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel A Casarotto, PhD, Principal Investigator — São Paulo University

IPD SHARING:
Plan to Share IPD: No